CLINICAL TRIAL: NCT00130039
Title: Trial for Efficacy and Safety of Cilostazol on the Progression of Symptomatic Intracranial Stenosis Comparing Clopidogrel
Brief Title: Trial of Cilostazol in Symptomatic Intracranial Arterial Stenosis II
Acronym: TOSS-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Korea Otsuka International Asia Arab (Industry)
Responsible Party: Sun U. Kwon, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TOSS-2
Record Dates: First submitted 2005-08-11; First posted 2005-08-15 (Estimated); Results first posted 2010-01-01 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2009-11

CONDITIONS: Cerebral Infarction; Atherosclerosis
Keywords: Infarction, Cerebral; cilostazol; stenosis; atherosclerosis; clopidogrel
MeSH Terms: conditions — Cerebral Infarction; Atherosclerosis; Constriction, Pathologic | interventions — Clopidogrel; Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cilostazol (Experimental): cilostazol 100mg bid plus placebo of clopidogrel
  Interventions: Drug: Cilostazol
- Clopidogrel (Active Comparator): clopidogrel 75mg qd and matching placebo of cilostazol
  Interventions: Drug: clopidogrel

INTERVENTIONS:
Drug: clopidogrel — Clopidogrel 75mg once a day plus placebo of cilostazol twice a day
  Other Names: Plavix, produced by Sanofi-Aventis.
  Arms: Clopidogrel
Drug: Cilostazol — Cilostazol 100mg twice a day plus placebo of clopidogrel once a day
  Other Names: cilostazol produced by Korea Otsuka Pharmaceutical
  Arms: cilostazol

SUMMARY:
This study will recruit 480 acute stroke patients with symptomatic intracranial stenosis (M1 segment of Middle cerebral artery (MCA) or basilar artery).

They will be randomly assigned into cilostazol group or clopidogrel group. Every patients will take 100mg of aspirin a day additionally.

The primary outcome variable of this study is Progression rate of symptomatic intracranial stenosis on magnetic resonance angiogram (MRA).

DETAILED DESCRIPTION:
[Goal] To Reveal the Effect and Safety of Cilostazol Compared with Clopidogrel on the Prevention of the Progression of Symptomatic Intracranial Arterial Stenosis.

[Trial Design] Double-Blind, Active-Controlled, Randomized, Multicenter Trial

[Participants] Acute ischemic stroke patients with symptomatic intracranial arterial stenosis

[Methods]

* Double-Blind, Active-Controlled, Randomized, Multicenter Trial
* Investigational product (Double Dummy Method):

Cilostazol 200mg (100mg twice per day) versus clopidogrel 75mg

* Concomitant medication: Aspirin 100 (75-150) mg per day
* Medication Duration: 7 months

[Outcome Variables]

Primary Outcome Variable:

* Progression rate of symptomatic intracranial arterial stenosis

Secondary outcome variables:

* The occurrence of new MRI (magnetic resonance image) lesion on follow-up MRI
* Stroke events
* Overall cardiovascular events: stroke, acute coronary syndrome, vascular death
* Ipsilateral ischemic stroke rate
* Fatal or major bleeding complications

ELIGIBILITY:
Inclusion Criteria:

* Cerebral infarction within 2 weeks from the onset or TIA with corresponding acute ischemic brain lesions on MRI within 2 weeks from the onset
* Age: more than 35 years of age
* Patient with significant focal stenosis in the M1 segment of middle cerebral artery (MCA) or basilar artery (BA) with acute ischemic lesions on magnetic resonance imaging (MRI) within the vascular territory of the stenosed artery.

Exclusion Criteria:

* Patients with any contraindications to the treatment with antiplatelet therapy
* Patients with potential cardiac embolic source; prosthetic valve, atrial fibrillation, atrial flutter, left atrial/atrial appendage thrombus, sick sinus syndrome, left ventricular thrombus, dilated cardiomyopathy, akinetic or hypokinetic left ventricular segment, atrial myxoma, Infective endocarditis, mitral valve stenosis or prolapse, mitral annuls calcification, left atrial turbulence, nonbacterial endocarditis, congestive heart failure, recent myocardial infarction (within 4 weeks)
* Patients with more than 50% stenosis in the parent artery of symptomatic stenosis
* Bleeding diathesis
* Chronic liver disease (ALT > 100 or AST > 100) or chronic renal disease (creatinine > 3.0mg/dl)
* Anemia (hemoglobin < 10mg/dl) or thrombocytopenia (platelet count less than 100,000/mm3)
* Nonatherosclerotic vasculopathy; patients with clinical characteristics suggesting arterial dissection, moyamoya disease, Takayasu's arteritis, radiation associated angiopathy, and other vasculitis.
* Severe stroke: NIH stroke scale : more than 16
* Pregnant or lactating patients
* Chronic user of NSAIDs
* Thrombolytic therapy for the symptomatic stenosis
* Symptomatic stenosis scheduled for angioplasty
* Patients with pacemaker or any other contraindications to MRI

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2005-08; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun U. Kwon, MD, PhD, Principal Investigator — Asan Medical Center, Univsersity of Ulsan, Medical College
Locations (19):
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Philippines (2):
  - Philippine General Hospital, Manila
  - University of Santo Tomas Hospital, Manila
- South Korea (13):
  - Konkuk Univ. Hospital, Seoul, Gwangjin-gu Hwayang-dong
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Dongguk University International Hospital, Goyang, Kyoungki-do
  - Hallym University Sacred Heart Hospital, Anyang, Kyunggi
  - Soonchunhyang University Hospital, Seoul, Seoul
  - Inha University Hospital, Inchon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Hallym University, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Boramae Hospital, Seoul
  - Eulji Hospital, Seoul
- Thailand (2):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok

REFERENCES:
- [Derived] Park TH, Lee JS, Park SS, Ko Y, Lee SJ, Lee KB, Lee J, Kang K, Park JM, Choi JC, Kim DE, Cho YJ, Kim JT, Kim DH, Cha JK, Han MK, Lee J, Oh MS, Yu KH, Lee BC, Bae HJ, Hong KS. Safety and efficacy of intravenous recombinant tissue plasminogen activator administered in the 3- to 4.5-hour window in Korea. J Stroke Cerebrovasc Dis. 2014 Aug;23(7):1805-12. doi: 10.1016/j.jstrokecerebrovasdis.2014.04.027. Epub 2014 Jun 21. PMID 24957314
- [Derived] Kim BJ, Rha JH, Kim SR, Kim DE, Kim HY, Lee JH, Bae HJ, Han MK, Kang DW, Ratanakorn D, Kim JS, Kwon SU. The effect of cilostazol on carotid intima-media thickness progression in patients with symptomatic intracranial atherosclerotic stenosis. J Stroke Cerebrovasc Dis. 2014 May-Jun;23(5):1164-70. doi: 10.1016/j.jstrokecerebrovasdis.2013.10.007. Epub 2013 Dec 6. PMID 24315720
- [Derived] Jung JM, Kang DW, Yu KH, Koo JS, Lee JH, Park JM, Hong KS, Cho YJ, Kim JS, Kwon SU; TOSS-2 Investigators. Predictors of recurrent stroke in patients with symptomatic intracranial arterial stenosis. Stroke. 2012 Oct;43(10):2785-7. doi: 10.1161/STROKEAHA.112.659185. Epub 2012 Aug 21. PMID 22910894
- [Derived] Kim DE, Kim JY, Jeong SW, Cho YJ, Park JM, Lee JH, Kang DW, Yu KH, Bae HJ, Hong KS, Koo JS, Lee SH, Lee BC, Han MK, Rha JH, Lee YS, Kim GM, Chae SL, Kim JS, Kwon SU. Association between changes in lipid profiles and progression of symptomatic intracranial atherosclerotic stenosis: a prospective multicenter study. Stroke. 2012 Jul;43(7):1824-30. doi: 10.1161/STROKEAHA.112.653659. Epub 2012 Apr 26. PMID 22539545
- [Derived] Kwon SU, Hong KS, Kang DW, Park JM, Lee JH, Cho YJ, Yu KH, Koo JS, Wong KS, Lee SH, Lee KB, Kim DE, Jeong SW, Bae HJ, Lee BC, Han MK, Rha JH, Kim HY, Mok VC, Lee YS, Kim GM, Suwanwela NC, Yun SC, Nah HW, Kim JS. Efficacy and safety of combination antiplatelet therapies in patients with symptomatic intracranial atherosclerotic stenosis. Stroke. 2011 Oct;42(10):2883-90. doi: 10.1161/STROKEAHA.110.609370. Epub 2011 Jul 28. PMID 21799173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 507 patients were registered www.toss2.com from 20 centers of 4 countries (Korea, Hongkong, Thailand, Philippines). 50 patients were excluded during case verification process because they did not satisfy patient's eligibility criteria.
  finally 457 patients were randomized into cilostazol or clopidogrel group
Pre-assignment Details: The excluded patients did not satisfy the definition of the symptomatic stenosis of our study protocol.
Groups:
- Cilostazol: cilostazol 100mg twice a day plus placebo of clopidogrel
- Clopidogrel: clopidogrel 75mg per day and matching placebo of cilostazol
Period: Overall Study
Arm/Group | Cilostazol | Clopidogrel
Started | 232 | 225
Completed | 202 (full analysis set) | 207 (full analysis set)
Not Completed | 30 | 18
Not completed — Withdrawal by Subject | 15 | 11
Not completed — Lost to Follow-up | 3 | 1
Not completed — Adverse Event | 4 | 2
Not completed — Physician Decision | 3 | 0
Not completed — clinical events without follow up MRI | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol | Clopidogrel | Total
Number analyzed (Participants) | 232 | 225 | 457
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 93 | 112 | 205
  >=65 years | 139 | 113 | 252
Age Continuous [Mean (Standard Deviation); unit: years] | 66.42 (11.33) | 64.58 (11.11) | 65.52 (11.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 113 | 223
  Male | 122 | 112 | 234
Region of Enrollment [Number; unit: participants]
  Philippines | 5 | 5 | 10
  Hong Kong | 11 | 12 | 23
  Thailand | 6 | 5 | 11
  Korea, Republic of | 210 | 203 | 413

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression of Symptomatic Intracranial Stenosis
Description: Blind reviewers classified the presence and severity of stenosis on middle cerebral arteries and basilar artery on magnetic resonance angiogram (MRA) into 5 grades; normal, mild, moderate, severe and occlusion. Progression was defined as worsening of stenosis by 1 or more grades on final MRA as compared with the baseline MRA.
  The progression of symptomatic stenosis is defined as 1 or more grade worsening of the stenosis on the symptomatic artery on MRA.
Time Frame: 7 months after treatment
Measure: Number; unit: participants
Arm/Group | Cilostazol | Clopidogrel
Number analyzed (Participants) | 202 | 207
participants | 20 | 32

2. Secondary Outcome: Number of Participants With New MRI (Magnetic Resonance Image) Lesions on Follow-up MRI
Description: number of patients with new ischemic lesions on FLAIR (Fluid attenuation inversion recovery) images of follow-up MRI, which were determined by slice to slice comparison with baseline MRI.
Time Frame: 7 months after treatment
Population: this analysis included the patients who had performed follow-up FLAIR imaging
Measure: Number; unit: pariticipants
Arm/Group | Cilostazol | Clopidogrel
Number analyzed (Participants) | 182 | 191
pariticipants | 34 | 23

3. Secondary Outcome: Number of Participants With Stroke Events
Description: including nonfatal ischemic stroke, nonfatal hemorrhagic stroke and fatal stroke
Time Frame: upto 7 months after randomization
Population: this outcome analysis performed on the intention to treat (ITT) method
Measure: Number; unit: participants
Arm/Group | Cilostazol | Clopidogrel
Number analyzed (Participants) | 232 | 225
participants | 11 | 7

4. Secondary Outcome: Number of Participants With Overall Cardiovascular Events
Description: including nonfatal stroke, nonfatal myocardial infarction and vascular death.
Time Frame: upto 7 months after randomization
Population: this outcome analysis was done intention to treat method
Measure: Number; unit: participants
Arm/Group | Cilostazol | Clopidogrel
Number analyzed (Participants) | 232 | 225
participants | 15 | 10

5. Secondary Outcome: Number of Patients With Ipsilateral Ischemic Stroke Rate
Description: ischemic stroke event which occured in the vascular territory of initial symptomatic stenosis
Time Frame: upto 7 months after randomization
Population: this outcome analysis was done ITT method
Measure: Number; unit: participants
Arm/Group | Cilostazol | Clopidogrel
Number analyzed (Participants) | 232 | 225
participants | 9 | 5

6. Secondary Outcome: Numbers of Fatal or Major Bleeding Complications
Description: life-threatening or fatal bleeding was defined as any fatal bleeding event, a drop in hemoglobin of ≥ 50g/L, or significant hypotension with need for inotropic agents, symptomatic intracranial hemorrhage, or transfusion of ≥ 4 units of red-blood cells or equivalent amount of whole blood. Major bleeding was defined as significantly disabling bleedings, intraocular bleeding leading to significant visual loss, or bleeding requiring transfusion of ≤ 3 units of red-blood cells or equivalent amount of whole blood
Time Frame: upto 7 months after randomization
Population: this outcome analysis was done ITT method
Measure: Number; unit: events
Arm/Group | Cilostazol | Clopidogrel
Number analyzed (Participants) | 232 | 225
events | 2 | 6

ADVERSE EVENTS:
Arm/Group | Cilostazol | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 54/232 | 54/225
Other Adverse Events (participants affected / at risk) | 232/232 | 225/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol (N=232) | Clopidogrel (N=225)
'Blood tinged loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
multi-organ failure (Infections and infestations) | 0 (0) | 1 (1)
abnormal involuntary movement (Nervous system disorders) | 1 (1) | 0 (0)
acute bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
acute myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3)
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
cerebral infarction (Nervous system disorders) | 10 (10) | 6 (6)
cerebral hemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
aneurysm unruptured (Vascular disorders) | 2 (2) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 5 (5) | 5 (5)
cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
GI bleeding (Gastrointestinal disorders) | 2 (2) | 6 (6)
traffic accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
cataract operation (Eye disorders) | 0 (0) | 3 (3)
depression (Psychiatric disorders) | 6 (6) | 4 (4)
diabetes complications (Endocrine disorders) | 2 (2) | 4 (4)
general weakness (Nervous system disorders) | 1 (1) | 3 (3)
vestibular neuronitis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
fracture or other joint pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (7)
infection (Infections and infestations) | 1 (1) | 2 (2)
headache (Nervous system disorders) | 3 (3) | 1 (1)
edema (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
seizure (Nervous system disorders) | 1 (1) | 0 (0)
severe hypertension (Cardiac disorders) | 1 (1) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cilostazol (N=232) | Clopidogrel (N=225)
headache (Nervous system disorders) | 62 (78) | 35 (42)
diarrhea (Gastrointestinal disorders) | 16 (18) | 9 (10)
petechia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
dizziness (Nervous system disorders) | 28 (29) | 21 (23)
palpitation (Cardiac disorders) | 7 (7) | 3 (3)
urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
epigastric soreness (Gastrointestinal disorders) | 15 (16) | 10 (10)
GI bleedings (Gastrointestinal disorders) | 3 (3) | 0 (0)
others (Social circumstances) | 169 (565) | 225 (564)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No